CLINICAL TRIAL: NCT04255173
Title: Anthropometric And Body Composition Measurements Related To Osteoporosis In Geriatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IMU OP
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Osteoporosis Senile; Obesity, Visceral
Keywords: osteoporosis; anthropometrics; body composition
MeSH Terms: conditions — Osteoporosis; Obesity, Abdominal | interventions — Body Mass Index; Waist Circumference; Body Height; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geriatric osteoporotic patients (Experimental): We measured different anthropometric and body composition measurements as body weight, BMI, percentage body fat, skeletal muscle index (SMI), ABSI, waist (WC) and hip circumference (HC) in geriatric population to investigate the relation to osteoporosis.
  Interventions: Diagnostic Test: Body mass index; Diagnostic Test: waist circumference; Diagnostic Test: hip circumference; Diagnostic Test: height; Diagnostic Test: Fat percentage; Diagnostic Test: Skeletal muscle index; Diagnostic Test: A body shape index (ABSI); Diagnostic Test: Dual energy x ray absorptiometry (DXA); Diagnostic Test: The Rapid Assessment of Physical Activity (RAPA) aerobic assessment

INTERVENTIONS:
Diagnostic Test: Body mass index — Body mass index is calculated as a ratio of height and weight, expressed as kg/m2
Diagnostic Test: waist circumference — waist circumference is measured as cm
Diagnostic Test: hip circumference — hip circumference is measured as cm
Diagnostic Test: height — height is measured as cm
Diagnostic Test: Fat percentage — Fat percentage and skeletal muscle mass (SMM) was calculated by using bioimpedance analysis (BIA) (Tanita TBF 300; Tanita Corp., Tokyo, Japan).
Diagnostic Test: Skeletal muscle index — Skeletal muscle index (SMI) was calculated from BIA-based skeletal muscle mass with a formula as SMM/height [m2].
Diagnostic Test: A body shape index (ABSI) — ABSI is measured as waist circumference (m) / (BMI(kg)2/3x Height(m)5/6)
Diagnostic Test: Dual energy x ray absorptiometry (DXA) — Osteoporosis is diagnosed with DXA scores. According to the T-scores calculated from femur neck (FN) and lumbar spine (LS), subjects divided into 3 groups as following: a) normal: T-score is greater than -1 SD (standard deviation), b) osteopenia: T-score is between -1 and -2.5 SD, c) osteoporosis: T-score is lower than -2.5 SD.
Diagnostic Test: The Rapid Assessment of Physical Activity (RAPA) aerobic assessment — Physical activity levels of patients were evaluated with The Rapid Assessment of Physical Activity (RAPA) aerobic assessment. Patients divided into 5 groups as following: 1 = sedentary, 2 = underactive, 3 = regular underactive (light activities), 4 = regular underactive, and 5 = regular active).

SUMMARY:
The patients who consulted to the geriatric outpatient clinic between 2018 and 2019 were included in the study. The inclusion criterions were being at or over the age of 65 and diagnosed with osteoporosis according to WHO criteria. Exclusion criteria include vertebral fracture due to known accidental traumas, history of drug therapy in the past year (biphosphonate, estrogen replacement therapy, glucocorticoids ), history of co-morbidities as malignancy, radiotherapy or chemotherapy, renal failure, hyperthyroidism, primer hyperparathyroidism, rheumatic disease or adrenal diseases.

Initially, a demographic form including age, sex, comorbidities, weight, height was filled by the participants. Body mass index (BMI, ratio of height and weight, expressed as kg/m2) calculated. Patients waist and hip circumference was measured (cm).

Fat percentage and skeletal muscle mass (SMM) was calculated by using bioimpedance analysis (BIA) (Tanita TBF 300; Tanita Corp., Tokyo, Japan). Skeletal muscle index (SMI) was calculated from BIA-based skeletal muscle mass with a formula as SMM/height [m2] [8]. ABSI is measured as waist circumference (m) / (BMI(kg)2/3x Height(m)5/6) [4].

Osteoporosis was evaluated by using dual energy x-ray absorptiometry (DXA). According to the T-scores calculated from femur neck (FN) and lumbar spine (LS), subjects divided into 3 groups as following: a) normal: T-score is greater than -1 SD, b) osteopenia: T-score is between -1 and -2.5 SD, c) osteoporosis: T-score is lower than -2.5 SD.

Physical activity levels of patients were evaluated with The Rapid Assessment of Physical Activity (RAPA) aerobic assessment [9]. Patients divided into 5 groups as following: 1 = sedentary, 2 = underactive, 3 = regular underactive (light activities), 4 = regular underactive, and 5 = regular active).

The study protocol was approved by the ethics committee (2018/0478) and all participants gave written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* being at or over the age of 65
* diagnosed with osteoporosis according to WHO criteria

Exclusion Criteria:

* vertebral fracture due to known accidental traumas
* history of drug therapy in the past year (biphosphonate, estrogen replacement therapy, glucocorticoids )
* history of co-morbidities as malignancy, radiotherapy or chemotherapy, renal failure, hyperthyroidism, primer hyperparathyroidism, rheumatic disease or adrenal diseases

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 571 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 2 years
  calculated as cm
Hip circumference | 2 years
  calculated as cm
Fat percentage | 2 years
  Fat percentage and skeletal muscle mass (SMM) was calculated by using bioimpedance analysis (BIA) (Tanita TBF 300; Tanita Corp., Tokyo, Japan)
Skeletal muscle index | 2 years
  Fat percentage and skeletal muscle mass (SMM) was calculated by using bioimpedance analysis (BIA) (Tanita TBF 300; Tanita Corp., Tokyo, Japan). Skeletal muscle index (SMI) was calculated from BIA-based skeletal muscle mass with a formula as SMM/height [m2]
A body shape index (ABSI) | 2 years
  ABSI is measured as waist circumference (m) / (BMI(kg)2/3x Height(m)5/6)

SECONDARY OUTCOMES:
The Rapid Assessment of Physical Activity (RAPA) aerobic assessment | 2 years
  Physical activity levels of patients were evaluated with The Rapid Assessment of Physical Activity (RAPA) aerobic assessment. Patients divided into 5 groups as following: 1 = sedentary, 2 = underactive, 3 = regular underactive (light activities), 4 = regular underactive, and 5 = regular active).

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Therapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No